CLINICAL TRIAL: NCT06537349
Title: Effects of 3% Diquafosol on Tear Film and Vision-related Quality of Life in Orthokeratology Lens Related Dry Eye
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DQS2024
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DQS group (Experimental): Participants in DQS group will be administered one drop of 3% DQS (Diquas, Santen Pharmaceutical Co.,Ltd., Osaka, Japan) six times per day for 4 weeks
  Interventions: Drug: 3% Diquafosol tetrasodium

INTERVENTIONS:
Drug: 3% Diquafosol tetrasodium — 3% Diquafosol tetrasodium eye drops will be used to assess its usefulness in OK lens related dry eye
  Other Names: Diquas

SUMMARY:
Investigate the effect of 3% Diquafosol on tear film and vision-related quality of life in dry eye patients wearing orthokeratology lenses(OK lens), and to provide reference for clinical treatment.This prospective, open label study will include 60 eyes of 30 OK lens related dry eye patients.Participants will receive 3% Diquafosol ophthalmic solution. The dosage for both drugs will be one drop, six times per day for 4 weeks. Pediatric Refractive Error Profiletear(PREP), tear film lipid layer (TFLL),non-invasive breakup time (NITBUT), corneoconjunctival staining score (CS), tear meniscus height (TMH), objective visual quality,ocular surface disease index (OSDI) will be assessed and compared at baseline, day-14, and day-28

DETAILED DESCRIPTION:
Keratoplasty is gaining popularity worldwide as a method of controlling myopia progression. Several clinical studies have shown that overnight wear of Orthokeratology lenses (OK) is an effective method of slowing myopia progression in adolescents.However, wearing corneal contact lenses tends to interfere with tear homeostasis, which may lead to ocular discomfort, dryness, and ocular surface disorders. More than 50% of contact lens wearers report symptoms of dry eye.Prolonged contact with the cornea can have an effect on the corneal layer.With the rapid increase in the use of OK lenses worldwide, potential complications have become a major concern for parents. Potential complications include keratitis and corneal epithelial damage. In addition, overnight OK lens wear has been associated with decreased tear production and reduced tear film stability. Recently, a four-week study by Carracedo et al. demonstrated that OK lens wear did not significantly change fluorescein-stained tear film breakup time or Schirmer's test I results, but subjects had increased dry eye symptoms one month after wear Decrease in cupped cell density.

Diquafosol Ophthalmic Solution (DQS) is a potent purinergic P2Y2 receptor agonist, a stabilized synthetic derivative of the naturally-occurring nucleotide uridine 5'-triphosphate; it stimulates the secretion of mucin and tears by conjunctival cup cells and conjunctival epithelial cells. Several studies have shown that Diquafosol sodium is effective in the treatment of dry eye. In addition, some studies have shown that Diquafosol sodium eye drops have significantly alleviated dry eye symptoms and improved ocular surface parameters in children wearing keratomileusis lenses at night. However, the available research lacks the ability of the DQS to assess the effect of DQS on visual acuity and quality of life improvement in patients with dry eye after wearing OK lenses. The results would inform clinicians to improve comfort and compliance with keratoplasty lenses in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years old
* Wearing corneal shape mirror more than one year and at least eight hours every night
* Myopia -5.50 to -1.00 D, astigmatism < 1.75 D, or curvature between 41.00 and 46.00D, astigmatism < -0.75D, and best corrected visual acuity ≥1.0.
* Diagnosis of dry eye: patients complained of dry eye, foreign body sensation, burning sensation, fatigue, discomfort, envy, subjective symptom such as vision fluctuation; (a) OSDI questionnaire score >13 points, and (b) NITBUT <10 s or (c) ocular surface dyeing assessment > 5 corneal spots/more than nine conjunctival spots.
* Participants were able to use eye drops as required, complete examinations, and return to the hospital for follow-up examinations within the specified time to complete follow-up.

Exclusion Criteria:

* Suffering from allergic or autoimmune disease associated with dry eye of the participants are not suitable for wearing OK lens
* Pathological changes in the corneal rim
* Eyelid rim lesions, cornea, uveitis, retina and other systemic diseases may affect the ocular surface. Examples include severe ocular surface diseases (Sjögren's syndrome, allergic conjunctivitis, ocular papules, conjunctival chafing, conjunctival scarring, and chemical damage);
* Received any dry eye treatment within 14 days prior to the start of this study or continued use of other topical eye drops that would affect the results of the study.
* Have received any other eye treatment or surgery

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Refractive Error Profile(PREP) questionnaire score | Day-0 (baseline), 2-weeks, 4-weeks
  Specifically to assess children's vision related quality of life, a total of 26 problem, original score for each from 5 points (positive) to 1 (negative), and then the original score for each minus 1 multiplied by 25, from 100 points (life quality) to 0 rating (poor quality of life), the average score for all 26 PREP problem of. "Strongly disagree" corresponds to 5 points when the statement is reversed.

SECONDARY OUTCOMES:
Non-invasive tear break-up time | Day-0 (baseline), 2-weeks, 4-weeks
  Changes in non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
Tear Film Lipid Layer | Day-0 (baseline), 2-weeks, 4-weeks
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
Conjunctivocorneal staining grade | Day-0 (baseline), 2-weeks, 4-weeks
  Using fluorescein sodium solution or fluorescein sodium test paper to contact the lower eyelid margin, corneal and conjunctival epithelial defects under the cobalt blue light of the slit lamp microscope showed different morphology, such as green spots, erosion, lamellar defects, ulcers and so on. The following categories: according to the severity of the symptoms can be mild, slit lamp microscope check no obvious signs of ocular surface damage (corneal fluorescein staining point < 5); Moderate: the extent of corneal damage under the slit lamp microscope did not exceed 2 quadrants and (or) the number of corneal fluorescein staining spots was >5 and <30. Severe: the range of corneal damage was 2 quadrants or more and (or) the corneal fluorescent staining spots were more than 30. The fluorescein staining spots in the cornea fused into thick spots, sheets or with filaments.
Tear meniscus height | Day-0 (baseline), 2-weeks, 4-weeks
  Changes in TMH will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
Ocular Surface Disease Index(OSDI) questionnaire score | Day-0 (baseline), 2-weeks, 4-weeks
  the Chinese language-validated OSDI, which is a questionnaire consisting of 12 questions for evaluating the effects of dry eye syndrome on vision, ocular symptoms, and any condition associated with DED, will be used. Te patient will answer each question on a scale ranging from 0 to 4, with 0 indicating "none of the time" and 4 indicating "all of the time." If a certain question is deemed irrelevant, it will be marked as "not applicable (N/A)" and excluded from the analysis. The OSDI total score is calculated according to the proprietary formula proposed by the authors of the original OSDI. The scale ranges from 0 to 100, with higher scores representing more severe cases of DED.
Objective visual quality assessment | Day-0 (baseline), 2-weeks, 4-weeks
  Using SCHWIND SIRIUS eyes analyzer objective visual quality assessment, including: total higher-order aberrations, spherical aberration, coma makes, clover, and RMS values etc..

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charm J, Cho P. High myopia-partial reduction ortho-k: a 2-year randomized study. Optom Vis Sci. 2013 Jun;90(6):530-9. doi: 10.1097/OPX.0b013e318293657d. PMID 23645372
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Kakita T, Hiraoka T, Oshika T. Influence of overnight orthokeratology on axial elongation in childhood myopia. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2170-4. doi: 10.1167/iovs.10-5485. PMID 21212181
- [Background] Chalmers RL, Young G, Kern J, Napier L, Hunt C. Soft Contact Lens-Related Symptoms in North America and the United Kingdom. Optom Vis Sci. 2016 Aug;93(8):836-47. doi: 10.1097/OPX.0000000000000927. PMID 27391535
- [Background] Han X, Xu D, Ge W, Wang Z, Li X, Liu W. A Comparison of the Effects of Orthokeratology Lens, Medcall Lens, and Ordinary Frame Glasses on the Accommodative Response in Myopic Children. Eye Contact Lens. 2018 Jul;44(4):268-271. doi: 10.1097/ICL.0000000000000390. PMID 28617728
- [Background] Li J, Dong P, Liu H. Effect of Overnight Wear Orthokeratology Lenses on Corneal Shape and Tears. Eye Contact Lens. 2018 Sep;44(5):304-307. doi: 10.1097/ICL.0000000000000357. PMID 28060144
- [Background] Carracedo G, Martin-Gil A, Fonseca B, Pintor J. Effect of overnight orthokeratology on conjunctival goblet cells. Cont Lens Anterior Eye. 2016 Aug;39(4):266-9. doi: 10.1016/j.clae.2016.04.001. Epub 2016 Apr 13. PMID 27085466
- [Background] Li Y, Kuang K, Yerxa B, Wen Q, Rosskothen H, Fischbarg J. Rabbit conjunctival epithelium transports fluid, and P2Y2(2) receptor agonists stimulate Cl(-) and fluid secretion. Am J Physiol Cell Physiol. 2001 Aug;281(2):C595-602. doi: 10.1152/ajpcell.2001.281.2.C595. PMID 11443059
- [Background] Ishikawa S, Sasaki T, Maruyama T, Murayama K, Shinoda K. Effectiveness and Adherence of Dry Eye Patients Who Switched from Short- to Long-Acting Diquafosol Ophthalmic Solution. J Clin Med. 2023 Jul 5;12(13):4495. doi: 10.3390/jcm12134495. PMID 37445527
- [Background] Keating GM. Diquafosol ophthalmic solution 3 %: a review of its use in dry eye. Drugs. 2015 May;75(8):911-22. doi: 10.1007/s40265-015-0409-7. PMID 25968930
- [Background] Amano S, Inoue K. Effect of topical 3% diquafosol sodium on eyes with dry eye disease and meibomian gland dysfunction. Clin Ophthalmol. 2017 Sep 14;11:1677-1682. doi: 10.2147/OPTH.S148167. eCollection 2017. PMID 29075094
- [Background] Ji YW, Kim HM, Ryu SY, Oh JW, Yeo A, Choi CY, Kim MJ, Song JS, Kim HS, Seo KY, Kim KP, Lee HK. Changes in Human Tear Proteome Following Topical Treatment of Dry Eye Disease: Cyclosporine A Versus Diquafosol Tetrasodium. Invest Ophthalmol Vis Sci. 2019 Dec 2;60(15):5035-5044. doi: 10.1167/iovs.19-27872. PMID 31800960
- [Background] Kaido M, Kawashima M, Shigeno Y, Yamada Y, Tsubota K. Randomized Controlled Study to Investigate the Effect of Topical Diquafosol Tetrasodium on Corneal Sensitivity in Short Tear Break-Up Time Dry Eye. Adv Ther. 2018 May;35(5):697-706. doi: 10.1007/s12325-018-0685-1. Epub 2018 Apr 18. PMID 29671255
- [Background] Yang Y, Wu Q, Tang Y, Wu H, Luo Z, Gao W, Hu Z, Hou L, Wang M, Yang Z, Li X. Short-term application of diquafosol ophthalmic solution benefits children with dry eye wearing orthokeratology lens. Front Med (Lausanne). 2023 Jul 13;10:1130117. doi: 10.3389/fmed.2023.1130117. eCollection 2023. PMID 37521335